CLINICAL TRIAL: NCT00501176
Title: Randomized Study Comparing the Effect of Plastic Stents to That of Expandable Metal Stents Prior to Pancreaticoduodenectomy
Brief Title: Preoperative Stent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ¨2006/220-31/4
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Pancreas Cancer
Keywords: Pancreas; cancer; SEMS; Plastic; stent; Whipple; Jaundicie
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Plastics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plastic stent (Active Comparator): Stent insertion
  Interventions: Procedure: Plastic and metalic stent inserion
- metalic stent (Active Comparator): Stent inserttion
  Interventions: Procedure: Plastic and metalic stent inserion

INTERVENTIONS:
Procedure: Plastic and metalic stent inserion — Patient randomizes to metal or plastic insertion prior to Whipple procedure
  Other Names: Two types of Stent prior to Whipple procedure

SUMMARY:
Randomized study comparing the effect of plastic stents to that of expandable metal stents as pre-operative drainage of the bile ducts prior to Whipple operation.

DETAILED DESCRIPTION:
Patients suffering from a locally invasive tumour process in the Periampullary area usually seek medical attention because of jaundice. Not only do patients suffering from jaundice show significant symptoms of exhaustion and purities, but they are also at higher risk for developing post-operative complications. Experimentally, the liver exhibits a reduced capacity for tolerating ischemia in the presence of jaundice. Several different etiologic factors suggest cause complication such as presence of toxic substances as bilirubin and bile salts, impaired nutritional status, effects of endotoxins, bacterial translocation, modulation of the inflammatory cascade with cytokine release, reduction of cellular immunity and nutritional. These complications primarily consist of septic complications (cholangitis, abscesses, and leakage), haemorrhage, impaired wound healing and renal disorders. Summarily, these issues have motivated pre-operative bile flow drainage by way of stent. Traditionally, pre-operative bile flow drainage has been achieved by insertion of a EP because these are considered easy to remove and cause less tissue reaction in the bile ducts. However, multiple studies have found the disadvantage with the EP is that it provides poorer bile drainage than the SEMS.

In palliative situations, metal stents have been associated with fewer side-effects in the form of fever relapse of jaundice, etc. These effects are likely due to better bile flow through the stent. It remains unclear if metal stents can provide similar advantages in the curative situation.

ELIGIBILITY:
Inclusion Criteria:

* The primary inclusion criteria are all patients with operable Periampullary cancer and jaundice who have not previously undergone bile flow drainage.

Exclusion Criteria:

* Define as failed ERCP, patients who have previously undergone bile flow drainage or radical surgery is not possible.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-12; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intra-operative measurement of the Culture from the bile. | Intraoperativt

SECONDARY OUTCOMES:
Intraoperative measurements of inflammatory reaction in the liver, hepatoduodenal ligament and around the bile ducts with biopsies. Stent dysfunction and cholangitis after ERCP and pre-operative bile flow relief. Postoperative analysis. | Perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Lars Enochsson, MD, PhD, Principal Investigator — Karolinksa Institutet; Urban Arnelo, M.D., Study Director — Karolinska Institutet; Lars Lundell, Professor, Study Chair — Karolinska Institutet
Locations (1):
- Karolinksa University Hospital, Stockholm, Sweden